CLINICAL TRIAL: NCT00078793
Title: Phase IV Registry of Etanercept (Enbrel®) In Children With Juvenile Rheumatoid Arthritis
Brief Title: Registry of Etanercept (Enbrel®) In Children With Juvenile Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Collaborators: Immunex Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 20021626; 016.0026; NCT00016575 (obsolete NCT alias)
Record Dates: First submitted 2004-03-05; First posted 2004-03-09 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Juvenile Rheumatoid Arthritis
Keywords: JRA; Registry
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Methotrexate group: Includes subjects being treated with methotrexate alone or in combination with other DMARDs with the exception of etanercept.
  Interventions: Drug: Enbrel®

INTERVENTIONS:
Drug: Enbrel® — Etanercept alone, etanercept plus methotrexate or other DMARDs

SUMMARY:
This study will evaluate long-term safety of etanercept with or without other DMARDs in children with polyarticular course or systemic juvenile rheumatoid arthritis (JRA) compared to a cohort of subjects with polyarticular or systemic JRA receiving methotrexate with or without other DMARDs.

ELIGIBILITY:
* JRA by American College of Rheumatology (ACR) criteria - Active joints - Initiate etanercept alone, etanercept plus methotrexate or other DMARDs, methotrexate alone, or methotrexate with other DMARDs within 6 months of entry into Registry
* Polyarticular or systemic RA in 3 or more joints at start of treatment

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric subjects age 2 to < or = 18 years of age with polyarticular course or systemic JRA who have recently started and are currently receiving: etanercept alone or in combination with methotrexate or other DMARDs; methotrexate alone or in combination with other DMARDs.The population includes pediatric subjects who completed Immunex protocol 016.0028 and selected other Immunex protocols will be eligible for this study once they change to marketed etanercept.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2000-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Adverse event rates and severity | 36 months of observation

SECONDARY OUTCOMES:
Growth data and Tanner scores | 36 months of observation

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Giannini EH, Ilowite NT, Lovell DJ, Wallace CA, Rabinovich CE, Reiff A, Higgins G, Gottlieb B, Chon Y, Zhang N, Baumgartner SW. Effects of long-term etanercept treatment on growth in children with selected categories of juvenile idiopathic arthritis. Arthritis Rheum. 2010 Nov;62(11):3259-64. doi: 10.1002/art.27682. PMID 20669280
- [Result] Giannini EH, Ilowite NT, Lovell DJ, Wallace CA, Rabinovich CE, Reiff A, Higgins G, Gottlieb B, Singer NG, Chon Y, Lin SL, Baumgartner SW; Pediatric Rheumatology Collaborative Study Group. Long-term safety and effectiveness of etanercept in children with selected categories of juvenile idiopathic arthritis. Arthritis Rheum. 2009 Sep;60(9):2794-804. doi: 10.1002/art.24777. PMID 19714630
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com